CLINICAL TRIAL: NCT05147675
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cells for the Treatment of Osteoarthritis
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cells for OA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-1-MSC-011
Record Dates: First submitted 2021-11-29; First posted 2021-12-07 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis; Spinal Arthritis
Keywords: Osteoarthritis; stem cell treatment; Spinal Arthritis
MeSH Terms: conditions — Osteoarthritis; Spondylarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloRx) (Experimental): Intravenous infusion and intraarticular injection (total dose of 100 million cells)
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of cultured allogeneic adult umbilical cord derived mesenchymal stem cells delivered intravenously and intraarticularly for the treatment of Osteoarthritis.

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of Osteoarthritis (OA). This patient funded trial aims to study the safety and efficacy of cultured allogeneic adult umbilical cord derived mesenchymal stem cells (UC-MSCs) for the treatment of OA. Patients with OA will receive intravenous infusion and intraarticular injection of UC-MSCs. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Osteoarthritis
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: Single Assessment Numeric Evaluation Score (SANE) | Four year follow-up
  ranging from 0 to 100%

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Athens Beverly Hills Medical Group, Glyfada, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Jin W, Liu H, Cui Y, Mao Q, Fei Z, Xiang C. [CURATIVE EFFECT OF HUMAN UMBILICAL CORD MESENCHYMAL STEM CELLS BY INTRA-ARTICULAR INJECTION FOR DEGENERATIVE KNEE OSTEOARTHRITIS]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2016 Dec 8;30(12):1472-1477. doi: 10.7507/1002-1892.20160305. Chinese. PMID 29786336
- [Background] Khalifeh Soltani S, Forogh B, Ahmadbeigi N, Hadizadeh Kharazi H, Fallahzadeh K, Kashani L, Karami M, Kheyrollah Y, Vasei M. Safety and efficacy of allogenic placental mesenchymal stem cells for treating knee osteoarthritis: a pilot study. Cytotherapy. 2019 Jan;21(1):54-63. doi: 10.1016/j.jcyt.2018.11.003. Epub 2018 Dec 3. PMID 30522806
- [Background] Zhao X, Ruan J, Tang H, Li J, Shi Y, Li M, Li S, Xu C, Lu Q, Dai C. Multi-compositional MRI evaluation of repair cartilage in knee osteoarthritis with treatment of allogeneic human adipose-derived mesenchymal progenitor cells. Stem Cell Res Ther. 2019 Oct 21;10(1):308. doi: 10.1186/s13287-019-1406-7. PMID 31639063
- [Background] Pers YM, Rackwitz L, Ferreira R, Pullig O, Delfour C, Barry F, Sensebe L, Casteilla L, Fleury S, Bourin P, Noel D, Canovas F, Cyteval C, Lisignoli G, Schrauth J, Haddad D, Domergue S, Noeth U, Jorgensen C; ADIPOA Consortium. Adipose Mesenchymal Stromal Cell-Based Therapy for Severe Osteoarthritis of the Knee: A Phase I Dose-Escalation Trial. Stem Cells Transl Med. 2016 Jul;5(7):847-56. doi: 10.5966/sctm.2015-0245. Epub 2016 May 23. PMID 27217345